CLINICAL TRIAL: NCT05057832
Title: Determination of Ustekinumab Levels in Patients With Crohn's Disease: Use in Clinical Practice
Brief Title: Determination of Ustekinumab Levels in Patients With Crohn's Disease
Acronym: Ustekinumab
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-UST-2021-01
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients treated with Ustekinumab.

SUMMARY:
Observational, prospective, single-center follow-up study carried out with patients from the area of the Virgen de Macarena University Hospital, diagnosed with chronic kidney disease, who started treatment with ustekinumab.

DETAILED DESCRIPTION:
Prospective follow-up observational study carried out with patients from the Virgen de Macarena University Hospital, under treatment with ustekinumab in the induction and maintenance phase in order to determine the cut-off points of the ustekinumab levels between which a clinical remission is expected in patients with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years.
* Patients treated with ustekinumab in induction and maintenance phase.
* They must agree to participate in the clinical study, having previously signed the informed consent.

Exclusion Criteria:

* Any patient who does not meet the inclusion criteria previously described and / or who refuses to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with ustekinumab who have had their levels measured will be included.
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Determine breakpoints. | Up to 44 weeks.
  To determine the breakpoints for ustekinumab levels between which clinical remission is expected in patients with inflammatory bowel disease.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Arguelles Arlas, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen de Macarena, Seville, Spain